CLINICAL TRIAL: NCT03113266
Title: A Phase II, Open, Multi-center and Single Arm Study Investigating Safety and Efficacy of Recombinant Humanized Anti-PD-1 mAb for Injection in Patients With Locally Advanced or Metastatic Bladder Urothelial Carcinoma
Brief Title: Safety and Efficacy of Toripalimab for Patients With Locally Advanced or Metastatic Bladder Urothelial Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Junshi Bioscience Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Junshi-JS001-009
Record Dates: First submitted 2017-04-06; First posted 2017-04-13 (Actual); Last update posted 2020-09-30 (Actual); Status verified 2020-09

CONDITIONS: Bladder Urothelial Carcinoma
Keywords: anti-PD-1 monoclonal antibody; Metastatic; Advanced; Bladder Urothelial Carcinoma
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- humanized anti-PD-1monoclonal antibody (Experimental): humanized anti-PD-1 monoclonal antibody is to be injected intravenously 3mg/kg Q2w until disease progresses or unacceptable tolerability occurs
  Interventions: Biological: humanized anti-PD-1 monoclonal antibody toripalimab

INTERVENTIONS:
Biological: humanized anti-PD-1 monoclonal antibody toripalimab — humanized anti-PD-1 monoclonal antibody (JS001) is a programmed death-1 (PD-1) immune checkpoint inhibitor antibody, which selectively interferes with the combination of PD-1 with its ligands, PD-L1 and PD-L2, resulting in the activation of lymphocytes and elimination of malignancy theoretically.
  Other Names: JS001, TAB001

SUMMARY:
This is a multi-center, open-label, phase 2 study evaluating the humanized anti-PD-1 antibody JS001, as a monotherapy in patients with locally advanced or metastatic bladder urothelial carcinoma who have failed in routine systemic treatment.

DETAILED DESCRIPTION:
This is a multi-center, open-label, phase 2 study evaluating the humanized anti-PD-1 antibody JS001, as a monotherapy in patients with locally advanced or metastatic bladder urothelial carcinoma who have failed in routine systemic treatment.The implementation of study meet the GCP.370 patients will be enrolled in the study to evaluate the safety and efficacy of JS001.Patients are injected with JS001 with 3mg/kg every 2 weeks until disease progresses or unacceptable toxicity occurs.Response assessment is conducted by every 8 weeks in first year, every 12 weeks in second year and every 16 weeks in third year and beyond.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female aged 18 and older are eligible;
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1;
* Histologic diagnosis of locally advanced or metastatic bladder urothelial carcinoma, including the origin of renal pelvis, ureter, urinary tract;
* At least 1 measurable lesion (only 1 measurable lymph node lesion is excluded) (routine CT scan >=20mm, spiral CT scan >=10mm, no prior radiation to measurable lesions);
* Providing with tumor specimen (for testing the expression of PD -L1 and the infiltrating lymphocytes);
* Predicted survival >=3 months;
* Brain or meningeal metastases must be disposed with surgery or radiation, and be stable clinically for at least 3 months (prior systemic steroids was allowed, but concurrent administration of systemic steroids with the study drug is excluded).
* Screening laboratory values must meet the following criteria（within past 14 days）:

hemoglobin ≥ 9.0 g/dL; neutrophils ≥ 1500 cells/ µL; platelets ≥ 100 x 10^3/ µL; total bilirubin ≤ 1.5 x upper limit of normal (ULN); aspartic transaminase (AST) and alanine transaminase (ALT) ≤ 2.5 x ULN without, and ≤ 5 x ULN with hepatic metastasis; serum creatinine ≤1╳ULN，creatinine clearance >50ml/min (Cockcroft-Gault equation) INR, aPTT≤1.5 x ULN; Urine protein + 1 or less, if the urine protein > 1 +, need to collect 24 hours urinary protein determination, the total amount should be 1 gram or less

* Without systemic steroids within past 4 weeks
* Males or female of childbearing potential must: agree to use using a reliable form of contraception (eg, oral contraceptives, intrauterine device, control sex desire, double barrier method of condom and spermicidal) during the treatment period and for at least 12 months after the last dose of study drug.
* Must have read, understood, and provided written informed consent voluntarily. Willing to adhere to the study visit schedule and the prohibitions and restrictions specified in this protocol.

Exclusion Criteria:

* Prior treatment with anti-PD-1/PD-L1/PD-L2 antibody, including auxiliary treatment phase
* Hypersensitivity to recombinant humanized anti-PD-1 monoclonal Abm or its components
* Prior antitumor therapy (including corticosteroids and immunotherapy) or participation in other clinical trials within past 4 weeks, or have not recovered from toxicities since the last treatment;
* Pregnant or nursing;
* Positive tests for HIV, HCV, HBsAg or HBcAb with positive test for HBV DNA (>500IU/ml);
* HBsAg or HBcAb with positive test for HBV DNA (>500IU/ml)
* History with active tuberculosis;
* Patients with any active autoimmune disease or a documented history of autoimmune disease, or history of syndrome that required systemic steroids or immunosuppressive medications, such as hypophysitis, pneumonia, colitis, hepatitis, nephritis, hyperthyroidism or hypothyroidism;
* Severe, uncontrolled medical condition that would affect patients' compliance or obscure the interpretation of toxicity determination or adverse events, including active severe infection, uncontrolled diabetes, angiocardiopathy (heart failure > class II NYHA, heart block >II grade, myocardial infarction, unstable arrhythmia or unstable angina within past 6 months, cerebral infarction within past 3 months) or pulmonary disease ( interstitial pneumonia, obstructive pulmonary disease or symptomatic bronchospasm);
* Evidence with active CNS disease;
* Prior live vaccine therapy within past 4 weeks;
* Received allogeneic hematopoietic stem cell transplantation or solid organ transplantation;
* Prior major surgery within past 4 weeks (diagnostic surgery excluded);
* Psychiatric medicines abuse without withdrawal, or history of psychiatric illness;
* Associated with clinical symptoms or symptomatic treatment of pleural effusion or ascites;
* Prior malignancy active within the previous 5 years except for locally curable cancers that have been apparently cured, such as basal cell skin cancer or carcinoma in situ of the cervix.
* Underlying medical condition that, in the Investigator's opinion, would increase the risks of study drug administration or obscure the interpretation of toxicity determination or adverse events.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 370 (Estimated)
Dates: Start 2017-04-06 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) by RECIST 1.1 and irRECIST | 3 years
  The treatment effect of JS001 will be assessed using irRC and RECIST 1.1 to determine tumor response.

SECONDARY OUTCOMES:
Duration of response (DOR) by RECIST1.1 and irRECIST | 3 years
  The treatment effect of JS001 will be assessed using irRC and RECIST 1.1 to determine duration of response.
Progression free survival (PFS) by RECIST1.1 and irRECIST | 3 years
  The treatment effect of JS001 will be assessed using irRC and RECIST 1.1 to determine progression-free survival time.
Overall survival (OS) | 3 years
  The treatment effect of JS001 will be assessed using irRC and RECIST 1.1 to determine overall survival.
Immunogenicity of anti-PD-1 monoclonal antibody | 3 years
  To test immunogenicity of anti-PD-1 monoclonal antibody
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 3 years
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0

OTHER OUTCOMES:
Correlation analysis of PD-L1 expression of tumor by ORR | 3 years
  correlation analysis of PD-L1 expression of tumor and objective response rate
Correlation analysis of PD-L1 expression of tumor by Immunohistochemistry | 3 years
  to analyse PD-L1 expression of tumor by Immunohistochemistry

CONTACTS AND LOCATIONS:
Overall Officials: Jun Guo, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes